CLINICAL TRIAL: NCT04717375
Title: A Phase 1/2, Dose Escalation, Dose Expansion, and Dose Optimization Study of the Safety, Tolerability, and Anti-tumor Activity of SAR444881 Administered Alone and in Combination With Pembrolizumab, Cetuximab and/or Chemotherapy in Participants With Advanced Solid Tumors
Brief Title: Study of SAR444881 Administered Alone and in Combination With Other Therapeutics in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCD17465; BND-22-001 (Other: Biond); U1111-1277-4421 (Other: WHO); 2023-504937-30-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; Cetuximab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SAR444881 Dose Escalation (Sub-Part 1A) (Experimental): Standard "3 + 3" dose escalation design with enrollment of at least 3 participants per dose level cohort. SAR444881 will be administered intravenously (IV), every 2 weeks (Q2W).
  Interventions: Drug: SAR444881
- SAR444881 in Combination with Pembrolizumab Dose Escalation (Sub-Part 1B) (Experimental): Standard "3 + 3" dose escalation design with enrollment of at least 3 participants per dose level cohort. SAR444881 and pembrolizumab will be administered intravenously (IV), every 3 weeks (Q3W).
  Interventions: Drug: SAR444881; Drug: Pembrolizumab
- SAR444881 in Combination with Cetuximab Dose Escalation (Sub-Part 1C) (Experimental): Standard "3 + 3" dose escalation design with enrollment of at least 3 participants per dose level cohort. SAR444881 and cetuximab will be administered intravenously (IV), every 2 weeks (Q2W).
  Interventions: Drug: SAR444881; Drug: Cetuximab
- SAR444881 Dose Optimization (Sub-Part 2A) (Experimental): SAR444881 Dose Optimization in combination with pembrolizumab/carboplatin/pemetrexed, pembrolizumab, or cetuximab. The indication for the combination cohorts will be non-squamous non-small cell lung cancer (NSCLC), gastric cancer or gastro-esophageal junction adenocarcinoma (GC/GEJ), colorectal carcinoma (CRC) any RAS. Enrollment will start after the recommended dose(s) of SAR444881 have been determined based on data from Sub-Parts 1A, 1B, and 1C.
  Interventions: Drug: SAR444881; Drug: Pembrolizumab; Drug: Cetuximab; Drug: Carboplatin; Drug: Pemetrexed
- SAR444881 Dose Expansion (Sub-Part 2B) (Experimental): The indication for this monotherapy cohort is cholangiocarcinoma. Enrollment will be opened based on emerging data from the dose-escalation phase and combination optimization data.
  Interventions: Drug: SAR444881

INTERVENTIONS:
Drug: SAR444881 — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: BND-22
Drug: Pembrolizumab — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Arms: SAR444881 Dose Optimization (Sub-Part 2A); SAR444881 in Combination with Pembrolizumab Dose Escalation (Sub-Part 1B)
Drug: Cetuximab — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Arms: SAR444881 Dose Optimization (Sub-Part 2A); SAR444881 in Combination with Cetuximab Dose Escalation (Sub-Part 1C)
Drug: Carboplatin — Pharmaceutical form: Concentrate for solution for infusion; Route of administration: Intravenous
  Arms: SAR444881 Dose Optimization (Sub-Part 2A)
Drug: Pemetrexed — Pharmaceutical form: Powder for concentrate for solution for infusion or concentrate for solution for infusion; Route of administration: Intravenous
  Arms: SAR444881 Dose Optimization (Sub-Part 2A)

SUMMARY:
The study will enroll advanced cancer patients with unresectable or metastatic disease who are refractory to or are not candidates for standard approved therapy. The study will be comprised of two parts - a dose escalation phase (Part 1) and a dose optimization/expansion phase (Part 2). Part 1 is comprised of three sub-parts: SAR444881 administered alone (Sub-Part 1A), SAR444881 administered in combination with pembrolizumab (Sub-Part 1B), and SAR444881 administered in combination with cetuximab (Sub-Part 1C). Part 2 is composed of two sub-parts: a dose optimization part where up to two doses of SAR444881 per indication are administered in combination with pembrolizumab, cetuximab, and/or carboplatin and pemetrexed (Sub-Part 2A); and a dose expansion part where SAR444881 is administered alone (Sub-Part 2B). In Sub-Part 2A, a two-stage design will be implemented to conduct dose optimization for each indication with combination therapy- Stage 1 (Preliminary Assessment) and Stage 2 (Randomization). Study is non-randomized except Stage 2 of Sub-Part 2A which will use randomization.

DETAILED DESCRIPTION:
Estimated Study Duration:

Dose Escalation (Part 1): Approximately 34 months Dose Optimization/Expansion (Part 2): Approximately 28 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic disease who are refractory to or are not candidates for standard approved therapy
* Histologic confirmation of malignancy
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG) of 0 or 1
* Participants must have adequate organ function as defined by laboratory tests
* Part 1: Following tumor types: Breast cancer, cervical cancer, colorectal cancer, adenocarcinoma or squamous cell carcinoma of the esophagus, gastric or gastroesophageal junction adenocarcinoma, squamous cell carcinoma of the head and neck, hepatobiliary cancers (hepatocellular carcinoma (HCC), gallbladder cancer, cholangiocarcinoma), non-small cell lung cancer, renal cell carcinoma, squamous cell carcinoma of the skin, pancreatic adenocarcinoma, ovarian cancer or urothelial carcinoma
* Part 2: Following tumor types: Squamous cell carcinoma of the head and neck, Gastric or gastroesophageal junction adenocarcinoma, non-squamous non-small cell lung cancer, non-small cell lung cancer, colorectal carcinoma (CRC) any RAS, and/or Cholangiocarcinoma

Exclusion Criteria:

* Active, known or suspected autoimmune disease
* Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Brain or leptomeningeal metastases
* Known history of positive test for HIV
* Non-HCC patients: acute or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV); HCC patients: untreated active HBV or dual infection with HBV/HCV
* Participants after solid organ or allogeneic hematopoietic stem cell transplant
* History of life-threatening toxicity related to prior immune therapy
* History of life-threatening toxicity related to prior cetuximab or other anti-EGFR antibodies (for Sub-Part 1C)
* Unstable or deteriorating cardiovascular disease within the previous 6 months
* Any major surgery within 4 weeks of study drug administration
* Prior/Concomitant Therapy:
* Cytotoxic/Non-cytotoxic anti-cancer agents, unless at least 4 weeks have elapsed from last dose
* Use of other investigational drugs within 28 days
* Prior treatment with macrophage or natural killer (NK) cells activating therapies
* Administration of a live attenuated vaccine within 28 days

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-04-11 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Part 1: Incidence of treatment-emergent adverse events (TEAEs) dose limiting toxicities (DLT) | Cycle 1 (28 days)
  Incidence of TEAEs meeting protocol defined DLT criteria
Part 1: Incidence of treatment-emergent adverse events and serious adverse events | Through study completion, an average of 5 months
Part 2: Objective Response Rate (ORR) per RECIST v1.1 | Through study completion, an average of 3 months
  Proportion of participants with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
Part 1: Objective Response Rate (ORR) per RECIST v1.1 | Through study completion, an average of 3 months
  Proportion of participants with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1
Part 1: Maximum observed plasma concentration [Cmax] | Through study completion, an average of 2 months
Part 1: Serum concentration at the end of the dosing interval (Ctrough) | Through study completion, an average of 2 months
Part 1: time of maximum observed serum concentration (Tmax) | Through study completion, an average of 2 months
Part 1: Terminal elimination half-life [T1/2] | Through study completion, an average of 2 months
Part 1: Area under the plasma concentration-time curve [AUC] | Through study completion, an average of 2 months
Part 1: Incidence of anti-drug antibodies (ADA) | Through study completion, an average of 5 months
Part 2: Progression Free Survival (PFS) | Up to 24 months
  Time from the date of first dose of study drug to the date of first documented disease progression or death due to any cause, whichever occurs first.
PFS rate | At 3, 6, 9, and 12 months, and up to 24 months
  Percentage of participants with PFS, per RECIST v1.1
Part 2: Duration of Response | Through study completion, an average of 6 months
  Duration between first documentation of CR or PR to first documentation of disease progression or death due to any cause, whichever occurs first
Part 2: Incidence of treatment-emergent adverse events and Serious Adverse Events | Through study completion, an average of 6 months
Part 2: Cmax | Through study completion, an average of 3 months
Part 2: Ctrough | Through study completion, an average of 3 months
Part 2: Tmax | Through study completion, an average of 3 months
Part 2: T1/2 | Through study completion, an average of 3 months
Part 2: AUC | Through study completion, an average of 3 months
Part 2: Incidence of ADA | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (18):
- United States (9):
  - Mayo Clinic Hospital- Site Number : 8400003, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center- Site Number : 8400002, Duarte, California
  - University of Colorado- Site Number : 8400012, Aurora, Colorado
  - Smilow Cancer Center at Yale-New Haven- Site Number : 8400001, New Haven, Connecticut
  - Clermont Oncology Center- Site Number : 8400005, Clermont, Florida
  - Mid Florida Hematology and Oncology Center- Site Number : 8400006, Orange City, Florida
  - Mercy Cancer Center - MercyOne Richard Deming Cancer Center- Site Number : 8400011, Des Moines, Iowa
  - Norton Cancer Institute - Downtown Women's Cancer Center- Site Number : 8400004, Louisville, Kentucky
  - Mayo Clinic Hospital Rochester- Site Number : 8400007, Rochester, Minnesota
- Canada (2):
  - Investigational Site Number : 1240001, Barrie, Ontario
  - Investigational Site Number : 1240003, Sherbrooke, Quebec
- Israel (5):
  - Investigational Site Number : 3760004, Haifa
  - Investigational Site Number : 3760005, Jerusalem
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760003, Ramat Gan
  - Investigational Site Number : 3760002, Tel Aviv
- United Kingdom (2):
  - Investigational Site Number : 8260003, London, London, City of
  - Investigational Site Number : 8260002, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Mandel I, Haves Ziv D, Goldshtein I, Peretz T, Alishekevitz D, Fridman Dror A, Hakim M, Hashmueli S, Friedman I, Sapir Y, Greco R, Qu H, Nestle F, Wiederschain D, Pao L, Sharma S, Ben Moshe T. BND-22, a first-in-class humanized ILT2-blocking antibody, promotes antitumor immunity and tumor regression. J Immunother Cancer. 2022 Sep;10(9):e004859. doi: 10.1136/jitc-2022-004859. PMID 36096532